CLINICAL TRIAL: NCT00945997
Title: Mifepristone (RU 486) and Misoprostol for Second Trimester Termination of Pregnancy. A Comparison of Two Different Dose Regimens.
Brief Title: Misoprostol for Second Trimester Termination of Pregnancy
Acronym: MIMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: JFGM Brouns, Zaans medical center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00.0427L
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Termination of Pregnancy Second Trimester
Keywords: misoprostol; mifepristone; medical abortion; randomised controlled trial
MeSH Terms: interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: misoprostol
- B (Active Comparator)
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — mifepristone 200 mg followed by 200 µg misoprostol per vaginam 36- 48 hours later at 4 hourly intervals (with a maximum of 10 administrations in 48 hours) until the foetus was delivered.
  Other Names: migegyne; cytotec
  Arms: A
Drug: misoprostol — mifepristone 200 mg followed by 400 µg misoprostol per vaginam 36- 48 hours later at 4 hourly intervals (with a maximum of 10 administrations in 48 hours) until the foetus was delivered.
  Other Names: mifegyne; cytotec
  Arms: B

SUMMARY:
To compare the efficacy of two different dose regimens of misoprostol administered vaginally in combination with mifepristone in second trimester termination of (non)viable pregnancy.

DETAILED DESCRIPTION:
The study was designed as a prospective double blinded randomised controlled trial, comparing 200µg to 400 µg misoprostol given vaginally at four hour intervals, starting 36-48 hours after the oral administration of mifepristone 200 mg at a gestational age between 14 to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with a gestational age between 14 to 24 weeks, confirmed by ultrasound, requesting termination of pregnancy

Exclusion Criteria:

* No informed consent
* Mifepristone allergy
* Chronic adrenal gland failure
* Kidney failure
* Liver failure
* Chronic use of corticosteroids
* COPD not responsive to treatment
* Cardiovascular disease
* Glaucoma

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2000-10; Primary Completion 2004-09 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Expulsion rate and the number of incomplete abortions warranting surgical evacuation of retained products of conception. | 8 weeks

SECONDARY OUTCOMES:
time between the first administration of misoprostol to to delivery of the foetus | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands